CLINICAL TRIAL: NCT06443372
Title: Gingival Crevicular Fluid Levels of Apoptotic Regulatory Proteins Bax and Bcl-xl in Stage III Periodontitis
Brief Title: GCF Bax and Bcl-xl Levels in Periodontitis
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Assoc. Prof., Aydin Adnan Menderes University
Other Study IDs: Apoptosis
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis; Gingivitis; Periodontal Health
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontitis: Periodontitis group (n = 23, generalized stage III) had interproximal CAL≥5 mm, along with PD≥6 mm and RBL extending to the mid-third of the root or beyond at 30% of the teeth or more. CAL was not originated from endodontic lesions draining through the marginal periodontium, dental caries extending into the cervical areas of the teeth, trauma-related gingival recession or distal bone loss in 2nd molars owing to extractions of 3rd molars. They had ≤4 teeth lost due to periodontitis.
  Interventions: Other: Clinical periodontal measurements, GCF sampling
- Gingivitis: Gingivitis group (n = 26) exhibited PD was ≤3 mm and BOP was ≥30% in the entire mouth as well as no detectable interproximal CAL or RBL.
  Interventions: Other: Clinical periodontal measurements, GCF sampling
- Periodontal Health: Periodontally healthy controls (n = 26) had clinically healthy gingiva on intact periodontium with PD ≤3 mm and BOP <10% and without detectable interproximal CAL and RBL.
  Interventions: Other: Clinical periodontal measurements, GCF sampling

INTERVENTIONS:
Other: Clinical periodontal measurements, GCF sampling — Clinical periodontal measuements included PD, CAL, BOP (+/-), GI, and PI. Clinical recordings were performed at six points (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, and distopalatal) of all teeth, except the 3rd molars.
  GCF samples were obtained 1 day following the clinical measurements. GCF was sampled with paper strips from two deepest pockets in periodontitis group; the most inflamed sites with clinical signs of redness or edema in gingivitis group; and the sites without visible inflammation in periodontally healthy group. GCF and saliva samples were stored at -80 °C until further analysis.

SUMMARY:
Intrinsic apoptosis pathway plays a critical role in the host immune defense and inflammation and its dysregulation is involved in various chronic diseases. Bcl-2 protein family primarly mediates this mitochondrial pathway. This study aimed to investigate the pro-apoptotic Bax and anti-apoptotic Bcl-xl levels and their association with interleukin-22 (IL-22) and transforming growth factor-beta 1 (TGF-β1) in gingival crevicular fluid (GCF) of patients with periodontitis. In total 75 systemically healthy and non-smoker individuals consisting of stage III periodontitis (n=23), gingivitis (n=26), periodontally healthy (n=26) were enrolled. Whole-mouth clinical periodontal measurements were recorded. Bax, Bcl-xl, IL-22 and TGF-β1 levels in GCF were determined by ELISA. Data were analyzed using non-parametric statistical tests.

DETAILED DESCRIPTION:
According to the 2017 World Workshop on the Classification of Periodontal and Peri-implant Diseases and Conditions, participants were categorized into three groups:

I. Periodontitis group (n=23), II. Gingivitis group (n=26) III. Periodontally healthy group (n=26)

Clinical periodontal measurements included probing depth (PD), clinical attachment loss (CAL), the dichotomous scoring of bleeding on probing (BOP +/-), gingival index (GI), and plaque index (PI). All clinical parameters were recorded at six points (mesiobuccal, buccal, distobuccal, mesiopalatal/mesiolingual, palatal/lingual, and distopalatal/distolingual) per tooth, except the 3rd molars, by a single investigator (C.Ö.) using a manual periodontal probe.

The percentage of radiographic bone loss (RBL) at the interproximal sites were calculated on the digital panoramic radiographs as the ratio of the distance between bone level and the cemento-enamel junction to the length of the root.

GCF samples were obtained 1 day following the clinical periodontal measurements. GCF was collected from the buccal aspects of non-contiguous interproximal sites in two single-rooted teeth via steril paper strips. Fluid samples were obtained from two deepest pockets in periodontitis group and the most inflamed sites with clinical signs of redness or edema in gingivitis group. In the periodontally healthy groups, samples were taken from the sites without visible inflammation. All samples were stored at -80 °C until further analysis.

Measurements of Bax, Bcl-xl, IL-22, and TGF-β1 levels in GCF samples were performed by the commercially available enzyme-linked immunosorbent assay (ELISA) kits. GCF molecule levels were expressed as total amounts at two samples per 30 s.

A statistical software package was used for all data analyses. The distribution of clinical and biochemical data was checked by Shapiro-Wilk's normality test. Since the data were not normally distributed, the differences between study groups in clinical measurements and GCF levels of Bax, Bcl-xl, IL-22, and TGF-β1 were compared by the Kruskal-Wallis non-parametric test with the Dunn-Bonferroni post hoc method. Spearman rank correlation analysis was performed to evaluate the correlations of four protein levels in GCF with clinical parameters. p<0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* No history of smoking
* At least 18 natural teeth (excluding 3rd molars)

Exclusion Criteria:

* Being diagnosed with diabetes mellitus, rheumatoid arthritis, cardiovascular system diseases, endocrine, immunologic, and mucocutaneous disorders
* Use of antibiotics, antihypertensives immunosuppressive and anti-inflammatory drugs within the past 6 months and topical antiseptic solutions in the last 3 months
* Having periodontal treatment in the previous year
* Wearing removable partial dentures or orthodontic appliances
* Restorative and endodontic therapy requirements
* Pregnant or nursing women

Ages: 27 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective case-control study consecutively enrolled 75 individuals (36 males and 39 females; aged 27 to 48 years; mean age, 37.30 ± 5.10 years) from the Department of Periodontology, School of Dentistry, Aydın Adnan Menderes University, Aydın, Turkey, in the period from March 2019 to January 2020.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
GCF Bax levels | 24 hours after clinical periodontal measurements
  Total amounts (ng)
GCF Bcl-xl levles | 24 hours after clinical periodontal measurements
  Total amounts (ng)

SECONDARY OUTCOMES:
GCF IL-22 levels | 24 hours after clinical periodontal measurements
  Total amounts (ng)
GCF TGF-β1 levels | 24 hours after clinical periodontal measurements
  Total amounts (ng)

CONTACTS AND LOCATIONS:
Overall Officials: Beral Afacan, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University, Faculty of Dentistry, Department of Periodontology, Aydin, Turkey (Türkiye)